CLINICAL TRIAL: NCT00122018
Title: N-acetylcysteine and Fenoldopam Protect the Renal Function of Patients With Chronic Renal Insufficiency Undergoing Cardiac Surgery.
Brief Title: An Investigation of N-acetylcysteine and Fenoldopam as Renal Protection Agents for Cardiac Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Linda F. Barr, M.D. (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor-Investigator, Linda F. Barr, M.D., Primary Investigator, Pulmonary Critical Care Associates of Baltimore
Organization: Pulmonary Critical Care Associates of Baltimore (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: REPORT
Record Dates: First submitted 2005-07-14; First posted 2005-07-21 (Estimated); Last update posted 2014-11-07 (Estimated); Status verified 2014-11

CONDITIONS: Kidney Failure, Acute; Kidney Failure, Chronic; Cardiac Surgical Procedures
Keywords: Kidney failure; Cardiac Surgery; Fenoldopam; N-acetylcysteine
MeSH Terms: conditions — Acute Kidney Injury; Kidney Failure, Chronic; Renal Insufficiency | interventions — Acetylcysteine; Fenoldopam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- NAC (Experimental): N-acetylcysteine started day prior to surgery, continued through night of surgery
  Interventions: Drug: N-acetylcysteine
- fenoldopam (Experimental): fenoldopam started at surgery continued for 24 hours
  Interventions: Drug: fenoldopam
- NAC and fenoldopam (Experimental): Both N-acetylcysteine and fenoldopam as above
  Interventions: Drug: N-acetylcysteine; Drug: fenoldopam
- Control (Placebo Comparator): Placebo

INTERVENTIONS:
Drug: N-acetylcysteine
  Other Names: Mucomyst
  Arms: NAC; NAC and fenoldopam
Drug: fenoldopam
  Other Names: Corlopam
  Arms: NAC and fenoldopam; fenoldopam

SUMMARY:
Patients with abnormal kidney function are at increased risk for complications following heart surgery, including worsening kidney function possibly requiring dialysis, a prolonged stay in the critical care unit and hospital, and the increased risk of death. Prior attempts at kidney protection for heart surgery patients have had mixed results. Two medicines, fenoldopam and N-acetylcysteine, have been shown to protect kidney function in other circumstances that cause kidney stress. The purpose of this study is to determine whether these medications will help to maintain the function of diseased kidneys during heart surgery.

DETAILED DESCRIPTION:
This is a randomized, double-blinded, placebo-controlled trial to evaluate fenoldopam and N-acetylcysteine (NAC) individually, and together, as renal protective agents for patients with renal insufficiency undergoing heart surgery. Subjects have chronic renal insufficiency with creatinine clearance (CrCl) </= 40cc/min but not on pre-operative dialysis, and receive: NAC 600 mg by mouth (po) twice a day (bid) or placebo starting 24 hours pre-operative and continuing through the day of surgery; and/or fenoldopam 0.1 mcg/kg/min intravenous (IV) or saline placebo at anesthetic induction and continuing for 48 hours. Outcome data include: nadir, post-operative day 3 and post-operative day 14 CrCl, time to CrCl nadir, length of Intensive Care Unit (ICU) stay, length of post-operative hospital stay, hospital costs, mortality, and the need for hemodialysis. Intraoperative and post-operative pressor use is being monitored. The enrollment will include 80 patients (20 in each group).

ELIGIBILITY:
Inclusion Criteria:

* Chronic creatinine clearance </= 40cc/h
* Pre-operative cardiac surgery

Exclusion Criteria:

* Pre-operative ongoing dialysis
* Nausea and vomiting
* Uncontrolled glaucoma
* Allergy to metabisulfite
* Enrollment in another clinical study within 30 days
* Pregnancy
* Acute renal failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2002-05; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Length of post-operative hospital stay | 30-day
Length of post-operative critical care stay | 30-day
Creatinine clearance post-operative days 3, 14, and nadir | 14 day

SECONDARY OUTCOMES:
Days to post-operative creatinine clearance nadir | 14 day
Intraoperative and post-operative pressor use (pressor-hours) | 48 hour
Hospital costs | 30-day
Mortality | 30-day

CONTACTS AND LOCATIONS:
Overall Officials: Linda F Barr, MD, Principal Investigator — Pulmonary and Critical Care Assoc. of Baltimore

REFERENCES:
- [Result] Barr LF, Kolodner K. N-acetylcysteine and fenoldopam protect the renal function of patients with chronic renal insufficiency undergoing cardiac surgery. Crit Care Med. 2008 May;36(5):1427-35. doi: 10.1097/CCM.0b013e31816f48ba. PMID 18434903
- [Derived] Esezobor CI, Bhatt GC, Effa EE, Hodson EM. Fenoldopam for preventing and treating acute kidney injury. Cochrane Database Syst Rev. 2024 Nov 28;11(11):CD012905. doi: 10.1002/14651858.CD012905.pub2. PMID 39607014